CLINICAL TRIAL: NCT00085748
Title: A Randomized, 6-Week Double-Blind, Placebo-Controlled Study With an Optional 24-Week Open-Label Extension to Evaluate the Safety and Tolerability of Flexible Doses of Paliperidone Extended Release in the Treatment of Geriatric Patients With Schizophrenia
Brief Title: Safety Study With Paliperidone ER Extended-Release (ER) Tablets in Geriatric Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004381
Record Dates: First submitted 2004-06-14; First posted 2004-06-16 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-11

CONDITIONS: Schizophrenia
Keywords: schizophrenia; geriatric; elderly
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: paliperidone ER

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of flexible dosages of paliperidone ER as compared with placebo in patients with schizophrenia who are 65 years of age or older. The primary objective of the open-label extension is the long-term assessment of safety and tolerability of paliperidone ER in patients diagnosed with schizophrenia.

DETAILED DESCRIPTION:
Paliperidone is being developed as a new therapeutic agent for the treatment of schizophrenia. The ER formulation of paliperidone was developed to deliver paliperidone at a relatively constant rate over a 24-hour period to improve the tolerability profile and decrease the potential for orthostatic hypotension. Typically, elderly persons with schizophrenia respond well to antipsychotic drugs. However, medications should be administered cautiously and usually at lower starting dosages than those prescribed for younger patients, with care taken to balance efficacy and tolerability. Flexible dosages of paliperidone ER have been chosen for this study to better achieve this balance and more closely mimic clinical practice. This is a multicenter, double-blind (neither the patient nor the physician will know if placebo or drug is being given and at what dose), randomized (patients will be assigned to different treatment groups based solely on chance), placebo-controlled, parallel-arm study. The primary purpose of the study is to evaluate the safety and tolerability of flexible doses of paliperidone ER in patients with schizophrenia who are 65 years of age or older. The study consists of a screening phase of up to 5 days, a 6-week double-blind treatment phase, and an optional 24-week open-label treatment phase. For administrative purposes, the screening and the double-blind treatment phases are referred to as R076477-SCH-302 and the open-label treatment phase is named R076477-SCH-702. Patients will be randomly assigned to receive paliperidone ER or placebo. At the time patients enter the double-blind period, they must be hospitalized for a minimum of 14 full days. Those patients who receive paliperidone ER will start at a dosage of 6 mg taken daily, which may be titrated up to a maximum of 12 mg or down to a minimum of 3 mg daily based on the patient's safety and tolerability of the drug. Patients who complete the 6 weeks of double-blind treatment, or who finish at least 21 days of treatment and discontinue because of lack of efficacy, may enter the 24-week open label treatment phase. While patients are hospitalized, efficacy will be assessed twice during the first week and at the end of the second week. Efficacy will be evaluated throughout the 6-week double-blind phase by completion of the Positive and Negative Syndrome Scale (PANSS), Clinical Global Impression Scale - Severity (CGI-S), Personal and Social Performance Scale (PSP), Schizophrenia Quality of Life Scale, Revision 4 (SQLS-R4), and Sleep Visual Analog Scale (VAS) during the double-blind treatment phase. The efficacy variable will be measured by the change from baseline score for PANSS, CGI S, SQLS-R4, Sleep VAS, and PSP. Safety will be monitored throughout the study based on incidence of adverse events; measurement of extrapyramidal symptoms using 3 rating scales (Abnormal Involuntary Movement Scale [AIMS], Barnes Akathisia Rating Scale [BARS], Simpson-Angus Rating Scale [SAS]); measurement of vital signs (blood pressure, heart rate); electrocardiograms; and clinical laboratory tests. Double-blind phase: paliperidone ER will be flexibly dosed in the range 3 to 12 mg (3, 6, 9, or 12 mg/day) orally once a day or matching placebo, for 6 weeks.

Open-label phase: The starting dose is 6 mg/day for 7 days; thereafter, flexible oral dosage of paliperidone ER (3, 6, 9, or 12 mg/day) for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Double-Blind Phase: 65 years of age or older
* DSM-IV diagnosis of schizophrenia for at least 1 year
* total PANSS score at screening and baseline between 70 and 120, inclusive
* agrees to hospitalization for a minimum of 14 days and for the duration of the study, if clinically indicated
* Open-label treatment phase: completed 6 weeks of the double-blind treatment phase or finished at least 21 days of treatment and discontinued because of lack of efficacy.

Exclusion Criteria:

* DSM-IV Axis I diagnosis other than schizophrenia
* DSM-IV diagnosis of substance dependence within the 6 months before screening (nicotine and caffeine dependence are not exclusionary)
* history of tardive dyskinesia or neuroleptic malignant syndrome (NMS)
* history of any severe preexisting severe gastrointestinal narrowing (pathologic or iatrogenic)
* previous history of a lack of response (2 adequate trials) to any antipsychotic

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2004-08; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Dosages and duration of treatment; incidence of adverse events throughout study. Changes from baseline to end of study in laboratory values, vital signs, electrocardiograms, and AIMS, BARS, and SAS scale scores.

SECONDARY OUTCOMES:
The change from baseline score to end point score at each point of measurement for PANSS, PSP, CGI S, SQLS-R4, and Sleep VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Tzimos A, Samokhvalov V, Kramer M, Ford L, Gassmann-Mayer C, Lim P, Eerdekens M. Safety and tolerability of oral paliperidone extended-release tablets in elderly patients with schizophrenia: a double-blind, placebo-controlled study with six-month open-label extension. Am J Geriatr Psychiatry. 2008 Jan;16(1):31-43. doi: 10.1097/JGP.0b013e31815a3e7a. PMID 18165460
- See also: Safety Study With Paliperidone ER Extended-Release (ER) Tablets in Geriatric Patients With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=586&filename=CR004381_CSR.pdf